CLINICAL TRIAL: NCT06330155
Title: A Genetic Study for Alzheimer Dementia: Case-control Study
Status: Not yet recruiting | Type: Observational
Sponsor: MinYoung Kim, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, MinYoung Kim, MD, PhD, Sponsor-Investigator, Bundang CHA Hospital
Organization: Bundang CHA Hospital (Other)
Other Study IDs: 2024-01-032
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Alzheimer Dementia (AD)
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alzheimer's dementia patient and healthy subjects

SUMMARY:
The purpose of this study is to find out the difference in genetic test results between Alzheimer's dementia patients and healthy subjects.

The investigators want to identify genes that are importantly related to Alzheimer's dementia.

ELIGIBILITY:
1. Inclusion Criteria: Alzheimer's dementia patient

   * Adult patients over 60 years old
   * Patients with a Alzheimer's dementia patient
   * Total Korean version of mini-mental state examination (K-MMSE) score less than 24
   * Total Clinical Dementia Rating (CDR) over 0.5
2. Inclusion Criteria: healthy subjects

   * Adult healthy over 60 years old
   * Total Korean version of mini-mental state examination (K-MMSE) over 24
   * Total Clinical Dementia Rating (CDR) is 0
3. Exclusion Criteria:

   * Those with severe medical conditions such as unstable conditions of the cardiovascular system, digestive system, respiratory system, endocrine system, etc., who are in poor general condition
   * In the case of a person with impaired consent (MMSE less than 10 points), if not accompanied by a guardian
   * Other cases where the researcher determines that participation in this clinical trial is not appropriate (Patients who are participating in other studies or have participated in other studies within the past 30 days can also participate in this study.)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10 Alzheimer's dementia patients 10 healthy subjects
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-03-26 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
genetic analysis | Baseline
  5cc blood collection for genetic testing

SECONDARY OUTCOMES:
Measurement of Korean version of mini-mental state examination (K-MMSE) | screening, Baseline
  K-MMSE is a measurement of cognitive level. Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe(≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment(MCI). The raw score may also need to be corrected for educational attainment and age.
Measurement of Clinical Dementia Rating (CDR) | screening, Baseline
  CDR is a rating scale for staging patients diagnosed with dementia. The CDR evaluates cognitive, behavioral and functional aspects of Alzheimer disease and other dementias. It is calculated on the basis of testing six different cognitive and behavioral domains such as memory, orientation, judgment and problem solving, community affairs, home and hobbies performance, and personal care. The CDR is based on a scale of 0-3: no dementia (CDR = 0), questionable dementia (CDR = 0.5), MCI (CDR = 1), moderate cognitive impairment (CDR = 2) and severe cognitive impairment (CDR = 3)
Measurement of Geriatric Depression Scale (GDSd) | Baseline
  GDS is a 30-item self-report assessment used to identify depression in the elderly. One point is assigned to each answer and the cumulative score is rated on a scoring grid. The grid sets a range of 0-9 as "normal", "10-19" as "mildly depressed", and 20-30 as "severely depressed".

CONTACTS AND LOCATIONS:
Overall Officials: MinYoung Kim, MD, PhD, Principal Investigator — CHA Bundang Medical Center